CLINICAL TRIAL: NCT02959385
Title: A Phase II Trial to Compare Efficacy and Safety of Definitive Radiochemotherapy VS Neoadjuvant Radiochemotherapy Plus Surgery in Patients Who Achieved Clinical Complete Response After Neoadjuvant Treatment for Stage II-III Esophageal Cancer
Brief Title: A Phase II Trial to Compare Efficacy and Safety of CRT VS Neo-CRT in Patients Who Achieved CCR for Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIH-PQS-2016090001
Record Dates: First submitted 2016-10-29; First posted 2016-11-09 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2016-10

CONDITIONS: Stage II Esophageal Cancer; Stage III Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Definitive Radiochemotherapy (Experimental): Concurrent Radiochemotherapy:
  Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day.
  Interventions: Radiation: Definitive Radiochemotherapy; Procedure: Neoadjuvant Radiochemotherapy
- Neoadjuvant Radiochemotherapy (Active Comparator): Concurrent Radiochemotherapy:
  Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.
  Interventions: Radiation: Definitive Radiochemotherapy; Procedure: Neoadjuvant Radiochemotherapy

INTERVENTIONS:
Radiation: Definitive Radiochemotherapy — Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day
Procedure: Neoadjuvant Radiochemotherapy — Concurrent Radiochemotherapy: Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.

SUMMARY:
Neoadjuvant chemoradiotherapy(Neo-CRT) plus surgery has been regarded as a standard of care for patients with resectable locally advanced oesophageal cancer. Many studies suggest that definitive Radiochemotherapy(CRT) has similar efficacy as neoadjuvant chemoradiotherapy plus surgery for esophageal cancers who respond to chemoradiation. Herein, a single center prospective randomized phase II clinical trial will be carried out to compare efficacy and safety of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection in patients who achieved clinical complete response(CCR) after neoadjuvant radiochemotherapy for stage II-III esophageal Cancer.

DETAILED DESCRIPTION:
1. Compare progression-free survival (PFS) and overall survival (OS) of definitive radiochemotherapy versus(VS) neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant treatment;
2. Compare the toxic and side effects of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete remission after neoadjuvant treatment;
3. Compare the relationship and consistency between pathological complete response of endoscopic biopsy specimens after neoadjuvant treatment and pathological complete response of surgical specimens in neoadjuvant radiochemotherapy plus radical resection group;
4. Assess impact of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection on quality of life of patients.

Clinical Complete Response After Neoadjuvant Treatment: Endoscope biopsy pathologic diagnosis indicate pathologic complete response after Neoadjuvant treatment; upper gastrointestinal/chest CT and symptom assessment indicate clinical complete response after Neoadjuvant treatment (Concurrent Radiochemotherapy: Radiotherapy, Intensity Modulation Radiation Therapy(IMRT), 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2), 1st/8th/15th/22nd day

ELIGIBILITY:
Inclusion Criteria:

1. Thoracic esophageal cancer patients or esophagocardial cancer patients, with locally advanced resectable tumor, clinically identified before treatment as T1-3N+M0 according to UICC(International Union Against Cancer) TNM(primary tumor, regional nodes, metastasis) Classification of Malignant Tumours, 7th ed.
2. Untreated patients who have not received any antitumor therapy
3. Life expectancy >6 months
4. Age: 18-70 years
5. White blood cell count ≥4.0×109/l, ANC(absolute neutrophil count) ≥1.5×109/l, thrombocyte count ≥1011/l, hemoglobin ≥90 g/l; normal liver and kidney functions
6. WHO PS(Performance Status): 0-1
7. Patients who understood the study and gave signed informed consent

Exclusion Criteria:

1. Patients who have already received antitumor therapy, including chemotherapy, radiotherapy or surgery;
2. Patients with hemorrhage or complicated hemorrhage
3. Other uncontrollable patients who are not suitable for surgery
4. Pregnant or lactating women
5. Patients who agree without acknowledgement as a result of psychological, family or social factors
6. Patients with CTCAE(Common Terminology Criteria Adverse Events Version 4.0) grade ≥2 peripheral neuropathy
7. Patients who have ever had malignant tumors other than esophageal cancer
8. Patients with a history of diabetes for >10 years with unsatisfactory control of blood glucose level
9. Patients with serious heart, lung, liver or kidney dysfunction, hematopathy, immune system disease or cachexia who therefore cannot tolerate chemotherapy or surgery
10. Others.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Compare overall survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Compare progression-free survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 years
  grade 3 or 4 toxicity of leukocytes, febrile neutropenia, thrombocytes, hemoglobin, nausea/vomiting, diarrhea, stomatitis, esophagitis, cardiovascular.
Comparison of pathological diagnosis between specimens of endoscopic biopsy and surgically resected in esophageal cancer | 2 years
  In the group of neoadjuvant radiochemotherapy plus surgery, we will compare the pathological diagnosis between specimens of endoscopic biopsy after neoadjuvant treatment and surgically resected.
Comparison between gross tumor volume (GTV) delineated with ultrasonic endoscopically placed titanium clips and GTV with conventional contouring method in thoracic esophageal cancer | 1 year
  patients undergo titanium clips placement on tumor boundaries under ultrasonic endoscopy before radiotherapy CT simulation. According to the clips, the reference GTVs are contoured by one experienced radiation oncologist. With the help of Eclipse treatment planning system, clips on CT are concealed. Two other radiation oncologists of expertise in oesophageal cancer delineate GTVs, defined as conventional GTVs, on the basis of endoscopy and oesophageal barium radiography. The two sets of GTVs are compared and analysed.
Determination of internal target volume (ITV) of thoracic esophageal cancer by evaluating movement of ultrasonic endoscopically placed titanium clips, with or without swallowing, during radiotherapy simulation | 1 year
  after titanium clips placement adjacent to esophageal cancer under ultrasonic endoscopy, clips movements in different borders and different directions are observed during radiotherapy simulation to determine the ITV of esophageal cancer, with or without swallowing.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsong Pang, Doctor, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian D, Chen X, Shang X, Wang Y, Tang P, Han D, Jiang H, Chen C, Zhao G, Zhou D, Cao F, Er P, Zhang W, Li X, Zhang T, Zhang B, Guan Y, Wang J, Yuan Z, Yu Z, Wang P, Pang Q. Definitive chemoradiotherapy versus neoadjuvant chemoradiotherapy followed by surgery in patients with locally advanced esophageal squamous cell carcinoma who achieved clinical complete response when induction chemoradiation finished: A phase II random. Radiother Oncol. 2022 Sep;174:1-7. doi: 10.1016/j.radonc.2022.06.015. Epub 2022 Jun 25. PMID 35764191